CLINICAL TRIAL: NCT06994299
Title: A Pilot Trial of Preoperative Irradiation With the STRIDE (Single Dose of Tremelimumab With Ongoing Durvalumab) Regimen (PRISM) for Resectable/Advanced Hepatocellular Carcinoma
Acronym: PRISM
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drug and financial support not available for the study.
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24-03027257
Record Dates: First submitted 2025-05-20; First posted 2025-05-29 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Hepatocellular Carcinoma (HCC)
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Radiotherapy; tremelimumab; durvalumab; Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Stereotactic Body Radiotherapy for HCC (Experimental): Hypofractionated radiotherapy - 8Gy x3 fractions (week 0) Tremelimumab - single dose of 300 mg IV (week 0). Durvalumab - 1500 mg IV every 4-weeks (weeks 0-3) prior to hepatic resection Surgery - hepatic resection (week 7)
  Interventions: Radiation: Radiation Therapy; Drug: Tremelimumab; Drug: Durvalumab; Procedure: Surgery

INTERVENTIONS:
Radiation: Radiation Therapy — Hypofractionated radiotherapy - 8Gy x3 fractions (week 0)
Drug: Tremelimumab — Tremelimumab - single dose of 300 mg IV (week 0).
Drug: Durvalumab — Durvalumab-500 mg IV every 4-weeks (weeks 0-3) prior to hepatic resection
Procedure: Surgery — Hepatic resection

SUMMARY:
This is an early-phase study testing a new combination treatment for cancer. participants will receive a type of radiation therapy called MRI-guided or CT-guided radiotherapy, depending on which imaging method is safe for them. The radiation will be given in three sessions, each delivering a moderate dose (8 Gray), focused only on the visible tumor.

At the same time, participants will receive immunotherapy, which is a treatment that helps the immune system fight cancer. This includes one dose of a drug called Tremelimumab and regular doses of another drug called Durvalumab, given every four weeks.

The goal of this study is to see if this combination is safe and shows signs of helping patients.

ELIGIBILITY:
Inclusion Criteria:

* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol. Written informed consent and any locally required authorization (e.g., Health Insurance Portability and Accountability Act in the US, European Union [EU] Data Privacy Directive in the EU) obtained from the patient/legal representative prior to performing any protocol-related procedures, including screening evaluations.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* Age ≥ 18 years
* ECOG performance status 0-1
* Life expectancy for at least 12 weeks
* Body weight >30kg
* LIRADS 5 or biopsy confirmed hepatocellular carcinoma (HCC)

  * Patients with histologically confirmed HCC (Documentation of original biopsy for diagnosis is acceptable if tumor tissue is unavailable) or clinical diagnosis by AASLD criteria in cirrhotic subjects is required (presence of arterial hypervascularity with venous washout).
  * For subjects without cirrhosis, histological confirmation is mandatory.
* Patient's must have resectable HCC. The determination of resectability status will ultimately lie in the clinical judgment of the surgical oncologist, medical oncologist, and radiation oncologist involved in the care of the patient.
* Patient must have measurable disease defined as a lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) and measures ≥ 15 mm with conventional techniques or

  o ≥ 10 mm with more sensitive techniques such as MRI or spiral CT (Computed Tomography) scan.
* Patient can have prior treatment for HCC including prior surgery, radiation therapy, local-regional therapy (ablation or arterial directed therapies), and systemic therapy including sorafenib or chemotherapy (but not anti-PD-1 or anti-CTLA-4 therapy).
* Patients with grade 2+ neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
* No evidence of distant metastases
* No infections requiring systemic antibiotic treatment
* Hgb >9.0 gm/dL, PLT > 100,000/mm3, total bilirubin ≤ 1.5x upper limit of normal

Exclusion Criteria

* Any other malignancy from which the patient has been disease-free for less than 5 years, except for non- melanoma skin cancer, or in situ carcinoma of any site.
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, and the laboratory values defined in the inclusion criteria
* Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab or tremelimumab may be included only after consultation with the Study Physician.
* Patients who have organ allografts.
* Patients who have had a major surgical procedure, open biopsy, or significant traumatic injury with poorly healed wound within 6 weeks prior to first dose of study drug; or anticipation of need for major surgical procedure during the study (other than defined by protocol); fine needle aspirations or core biopsies within 7 days prior to first dose of study drug. NOTE: Patients will be allowed to start cycle 1 day 1 therapy after 24 hours from pre-treatment biopsy.
* Autoimmune disease: Patients with a history of inflammatory bowel disease (including Crohn's disease and ulcerative colitis) are excluded from this study as are patients with a history of autoimmune disease (e.g., rheumatoid arthritis, systemic progressive sclerosis [scleroderma], systemic lupus erythematosus, autoimmune vasculitis [e.g., Wegener's granulomatosis]).
* Known history of testing positive for human immunodeficiency virus (HIV) (positive HIV 1 /2 antibodies) or known acquired immunodeficiency syndrome (AIDS).
* Active tuberculosis infection (clinical evaluation that may include history, physical examination, and radiographic findings or tuberculosis testing in line with local practive).
* Any underlying medical condition, which, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of adverse events, such as a condition associated with frequent diarrhea.
* Patients who have had a history of acute diverticulitis, abdominal fistula, gastrointestinal perforation, intra- abdominal abscess, GI obstruction, abdominal carcinomatosis which are known risks factors for bowel perforation, should be excluded from the study.Patients who have a primary brain tumor (excluding meningiomas and other benign lesions), any brain metastases, leptomeningeal disease, seizure disorders not controlled with standard medical therapy, or history of stroke within the past year.
* History of serious systemic disease, including myocardial infarction or unstable angina within the last 12 months, history of hypertensive crisis or hypertensive encephalopathy, uncontrolled hypertension (blood pressure of >140/90 mmHg) at the time of enrollment, New York Heart Association (NYHA) Grade II or greater congestive heart failure, unstable symptomatic arrhythmia requiring medication (patients with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), significant vascular disease or symptomatic peripheral vascular disease.
* Patients who have history of other diseases, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2027-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety, as measured by the number of Grade 3+ CTCAE treatment related toxicity rates within three months from start of treatment | Within 3 months from start of treatment
Efficacy, as measured by major pathologic response rates determined from resected surgical specimens | Week 7

SECONDARY OUTCOMES:
Feasibility as measured by the recruitment timeline | 24 months
  The desired requirement timeline is to enroll 10 participants in 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Encouse Golden, M.D.,PHD, Principal Investigator — Weill Cornell Medicine, New York, NY, USA
Locations (1):
- New York-Presbyterian Weill Cornell Medical College, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No